CLINICAL TRIAL: NCT01276535
Title: A Pilot Study to Evaluate the Efficacy of Low-level Laser Therapy in Reducing Blemishes by Quantifying a Decrease in Signs of Blemishes, Both Non-inflammatory and Inflammatory
Brief Title: Study of the Use of Low Level Laser Therapy to Reduce Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECACNEP1
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erchonia MLS + Erchonia THL (Experimental): The Erchonia® MLS contains 5 independent diodes: 4 each emitting 17 milliwatt (mW) 635 nanometers (nm) of red laser light and the fifth diode emitting 17 mW, 405 nm of blue laser light.
  The Erchonia THL is a single diode pulsed laser that emits 4.9 milliwatts (mW) of red 635 nanometer (nm) light.
  Interventions: Device: Erchonia MLS + Erchonia THL

INTERVENTIONS:
Device: Erchonia MLS + Erchonia THL — The Erchonia® MLS is administered weekly for 6 continuous weeks at the test site by the study investigator.
  The Erchonia THL is administered twice daily for 6 continuous weeks (42 days) at home by the subject.
  Administration of the MLS and the THL occur simultaneously over the 6-week administration phase.
  The intent is to evaluate the effectiveness of Erchonia MLS & Erchonia THL when administered together, and not to compare Erchonia MLS vs. Erchonia THL

SUMMARY:
The purpose of this study is to determine whether low level laser light therapy is effective in the treatment of acne blemishes.

DETAILED DESCRIPTION:
Acne is a chronic inflammatory disorder plaguing the sebaceous follicle, and debate still remains over what truly initiates lesion formation. Experts agree that an increase in androgen production plays a significant role in the onset of acne. Androgens promote the increase in size of sebaceous glands and stimulate sebum production. The simple act of sebaceous gland stimulation via androgens could ultimately promote the upregulation of pro-inflammatory cytokines like tumor necrosis factor-α (TNF-α) and interleukin (IL-1α) without propionibacteria even being present. The synthesis of IL-α and other pro-inflammatory cytokines including prostaglandins occurs via the inducible enzyme known as cyclooxygenase-2 (COX-2). Studies analyzing the pathogenesis of mucositis have identified COX-2 as an important contributor to the upregulation of pro-inflammatory cytokines and thus a major contributor to the progression of the disorder itself.

Recent evidence indicates that low-level laser therapy (LLLT) is able to significantly diminish the expression of COX-2, resulting in the reduction of inflammation. The ability to modulate the COX-2 pathways via LLLT is believed to inhibit the production of pro-inflammatory cytokines (i.e. TNF-α and IL- α) present in acne-prone skin.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent form.
* male or female.
* 18 to 40 years.
* area sought for acne reduction is the face.
* diagnosis of moderate or severe acne vulgaris, defined as grade 3-5 according to the grading criteria of acne severity given by Burton et al.
* Acne has been ongoing for at least 3 months prior to screening and must include inflammatory lesions.
* female using hormonal birth control must have been on a stable dose for at least 3 months prior to screening.
* negative pregnancy test for female subjects, unless the female subject has been surgically sterilized.
* sexually active female subject who is not surgically sterile or 2 years post menopausal must agree to use approved contraception/birth control measure while on study
* PI (A normal healthy patient) or P2 (A patient with mild systemic disease) on the American Society of Anesthesiologists (ASA) Physical Status Classification System.
* subject agrees to abstain from use of non-study treatments for acne while enrolled in the study.
* subject agrees to abstain from use of tanning beds/sunbathing while partaking in the study.
* subject agrees, and be able, to maintain regular medication schedule, as is medically feasible, during study participation.
* subject agrees to not change skin care regimen throughout study participation.
* subject is willing and able to comply with all requirements of the study protocol.

Exclusion Criteria:

* use of topical acne treatment within 15 days prior to start of study.
* use of oral acne treatment within 30 days prior to the start of study.
* use of oral isotretinoin or other systemic retinoids in the 12 months preceding the start of the study.
* use of systemic steroids within 30 days prior to the start of the study.
* pregnancy or currently nursing, or planning pregnancy during the course of the study
* participation in any clinical study involving an investigational product within 30 days of the start of the study
* use of tanning beds or sunbathing in the 30 days prior to the start of the study.
* history of keloids or other photosensitive disorders or use of any photosensitizing medication.
* currently taking any medication that may alleviate or exacerbate acne.
* Porphyria or known allergies to porphyrins.
* current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.
* known malignancy or history of malignancy other than non-melanoma skin cancer
* human immunodeficiency virus (HIV), hepatitis B or hepatitis C
* signs of bacterial, fungal or viral skin lesions that may interfere with assessment of acne vulgaris.
* known inherited or acquired coagulation defects.
* substance abuse (drug or alcohol) problem within the previous 3 years.
* developmental disability or cognitive impairment that may preclude study compliance.
* unlikely to comply with the study protocol and procedure administration protocol, or is considered unsuitable for participation in the study for any other reason in the opinion of the investigator.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Nikolaidis, MD, Principal Investigator
Locations (1):
- Westlake Dermatology, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 subjects were recruited and enrolled from March 2, 2010 through April 29, 2010 at one medical clinic.
Pre-assignment Details: There were no significant events or approaches for the overall study following participant enrollment, but prior to group assignment. There were no enrolled participants excluded from the trial before assignment to groups.
Groups:
- Erchonia MLS & Erchonia THL: The Erchonia® MLS contains 5 independent diodes: 4 that each emit 17 milliwatt (mW) 635 nm of red laser light and the fifth diode that emits 17 mW, 405 nm of blue laser light. The MLS is administered weekly for 6 continuous weeks at the test site by the study investigator.
  The Erchonia® THL is a single diode pulsed laser that emits 4.9 mW of red 635 nm light, The THL is administered twice daily for 6 continuous weeks (42 days) at home by the subject.
Period: Overall Study
Arm/Group | Erchonia MLS & Erchonia THL
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erchonia MLS & Erchonia THL
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (5.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Grade on the Burton et al. Acne Severity Grade Scale
Description: The Burton et al. Acne Severity Grade Scale grades the type of acne lesion from Grade 0: no acne lesions through Grade 1: sub-clinical acne, Grade 2: mild acne, Grade 3: moderate acne; Grade 4: severe acne, to Grade 5: extremely severe acne. The number of participants whose entire face demonstrated an improvement of one or more grades on the Burton et al. Acne Severity Scale at week 6 relative to baseline was calculated.
Time Frame: baseline and 6 weeks
Measure: Number; unit: participants
Arm/Group | Erchonia MLS & Erchonia THL
Number analyzed (Participants) | 12
participants | 2

2. Secondary Outcome: Change From Baseline in Inflammatory Lesion Count at 6 Weeks
Description: The number of pustules, papules and nodules are summed to attain a total inflammatory lesion count.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Erchonia MLS & Erchonia THL
Number analyzed (Participants) | 10
lesions | -9.75 (4.56)
Statistical Analysis 1: Comparison: Erchonia MLS & Erchonia THL; Comparison is made of the combined application of the Erchonia MLS and the Erchonia THL. Results are analyzed at 6 weeks relative to Baseline; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

3. Secondary Outcome: Change From Baseline in Non-Inflammatory Lesion Count at 6 Weeks
Description: The number of open comedones and closed comedones are summed to attain the total non-inflammatory lesion count.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Erchonia MLS & Erchonia THL
Number analyzed (Participants) | 12
lesions | -77.00 (21.78)
Statistical Analysis 1: Comparison: Erchonia MLS & Erchonia THL; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 weeks of treatment administration and 6 weeks of follow-up.
Arm/Group | Erchonia MLS & Erchonia THL
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No